CLINICAL TRIAL: NCT06136585
Title: Comparison of Efficacy of Sugammadex Versus Neostigmine in Reversing Neuromuscular Blocks in Patients Having Outpatient Endoscopic Retrograde Cholangiopancreatography (ERCP). A Randomized, Double-Blinded Trial
Brief Title: Sugammadex Vs Neostigmine in Reversing Neuromuscular Blocks in Outpatient ERCP. A Randomized, Double-Blinded Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ryu Komatsu, MD, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-378
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Neuromuscular Blocks
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: A single-center, Assessor-Blinded, parallel group randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2 mg/kg sugammadex (Experimental): All participants will be given rocuromium for neuromuscular blocks during the procedure. Per randomization, patients in this group will be reversed with 2 mg/kg sugammadex.
  Interventions: Drug: 2 mg/kg sugammadex
- 0.07 mg/kg neostigmine (Active Comparator): All participants will be given rocuromium for neuromuscular blocks during the procedure. Per randomization, patients in this group will be reversed with 0.07 mg/kg neostigmine (to a maximum of 5 mg).
  Interventions: Drug: 0.07 mg/kg neostigmine

INTERVENTIONS:
Drug: 2 mg/kg sugammadex — All participants will be given rocuromium for neuromuscular blocks during the procedure. Per randomization, patients in this group will be reversed with 2 mg/kg sugammadex.
  Other Names: All participants will be given rocuromium for neuromuscular blocks during the procedure. Per randomization, patients in this group will be reversed with 2 mg/kg sugammadex.
  Arms: 2 mg/kg sugammadex
Drug: 0.07 mg/kg neostigmine — All participants will be given rocuromium for neuromuscular blocks during the procedure. Per randomization, patients in this group will be reversed with 0.07 mg/kg neostigmine (to a maximum of 5 mg).
  Other Names: All participants will be given rocuromium for neuromuscular blocks during the procedure. Per randomization, patients in this group will be reversed with 0.07 mg/kg neostigmine (to a maximum of 5 mg).
  Arms: 0.07 mg/kg neostigmine

SUMMARY:
The investigators propose a single-center, assessor-Blinded, parallel group randomized trial to compare the efficacy of reversal of rocuronium induced neuromuscular blockade by sugammadex versus neostigmine in patients undergoing Endoscopic retrograde cholangiopancreatography at Cleveland Clinic Fairview Hospital.

DETAILED DESCRIPTION:
The investigators propose a single-center, assessor-blinded, parallel group randomized trial to compare the efficacy of reversal of rocuronium induced neuromuscular blockade by sugammadex versus neostigmine. Participating patients and outcome assessors will be blinded to group assignment. The anesthesiologists who assume anesthesia care will not be blinded to group assignment.

American Society of Anesthesiologists (ASA) physical status 3 and 4 adults scheduled for elective outpatient ERCP procedure with general anesthesia at Cleveland Clinic Fairview Hospital will be included in the study. Patients will be excluded if they have suspected difficult airway, neuromuscular disorders, end-stage renal disease requiring hemodialysis, are allergic to fentanyl, neuromuscular blocking drugs or neuromuscular reversal drugs, or are pregnant or breastfeeding.

Eighty patients scheduled for outpatient ERCP with general anesthesia and rocuronium-induced muscle relaxation will be randomized 1:1 to: 1) reversal by sugammadex; or 2) reversal by neostigmine. Randomization will be stratified by 2 factors: (1) patient's age (older than 60 versus younger than 60) and (2) diagnostic vs. interventional procedures. Randomization will be based on computer generated codes that will be maintained in web-based system until shortly before induction of anesthesia, thus concealing allocation so long as practical.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* American Society of Anesthesiologist physical status 3-4
* Scheduled for outpatient endoscopic retrograde cholangiopancreatography

Exclusion Criteria:

* Difficult Airway
* Neuromuscular Disorders (eg: ALS, Botulism, Myasthenia Gravis, Lambert-eaton syndrome)
* End stage renal disease requiring dialysis
* Pregnancy or breast-feeding
* Allergy to Fentanyl
* Allergy to Neuromuscular blocking drugs (eg: rocuronium)
* Allergy to Neuromuscular reversal drugs (eg: sugammadex or neostigmine)
* Allergy to glycopyrrolate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time required from reversal of neuromuscular block to discharge readiness | First 24 hours after reversal of neuromuscular block
  To assess the time required from reversal of neuromuscular block to discharge readiness in patients randomized to sugammadex or neostigmine.

SECONDARY OUTCOMES:
Incidence of postoperative nausea and vomiting (PONV) in patients randomized to sugammadex or neostigmine. | 2 hours of post anesthetic recovery
  Incidence of postoperative nausea and vomiting (PONV) in patients randomized to sugammadex or neostigmine.

CONTACTS AND LOCATIONS:
Overall Officials: Ryu Komatsu, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Fairview Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cotton PB. Are low-volume ERCPists a problem in the United States? A plea to examine and improve ERCP practice-NOW. Gastrointest Endosc. 2011 Jul;74(1):161-6. doi: 10.1016/j.gie.2011.03.1233. No abstract available. PMID 21704815